CLINICAL TRIAL: NCT04717401
Title: Strain-Counterstrain Versus Muscle Energy Technique In Sacroiliac Joint Dysfunction
Brief Title: Comparison Between Strain-counterstrain and Muscle Energy Technique in Sacroiliac Joint Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Karima Abdelaty Hassan, Lecturer of Physical Therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: sacroiliac dysfunction
Record Dates: First submitted 2021-01-01; First posted 2021-01-22 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Sacroiliac Joint Somatic Dysfunction
Keywords: Strain-counterstrain; Muscle energy technique

STUDY DESIGN:
Who Masked: Participant
Masking Description: The patients will be assigned randomly to the 2 groups by using opaque, sealed envelopes, containing the name of one of each groups (SCS or MET). A colleague who will be not participating in recruiting, treating or evaluating participants will select the envelopes. After the initial assessment but before the first therapy session, group allocation will be carried out.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strain-counterstrain Group A (Experimental): Strain Counterstrain (SCS) is a passive positional technique which aims to relieve musculoskeletal pain and dysfunction by indirect manipulation .
  Interventions: Procedure: Strain-Counterstrain
- Muscle Energy Technique Group B (Experimental): MET is a gentle manual therapy for the restricted mobility of the spine and extremities and is an active procedure in which the corrective force is regulated by the patient, not the clinician. This technique requires the patient to perform voluntary muscle contractions of varying intensity, in a specific direction, while the clinician uses a counter-force that does not allow movement to occur The physiological mechanism underlying SCS is unknown though. It has hypothesized that muscle tone inhibition occurs by stimulation of the target muscle's Golgi tendon organ by physical approximation of muscle origin and insertion.
  Interventions: Procedure: Muscle Energy Technique

INTERVENTIONS:
Procedure: Strain-Counterstrain — Strain-counterstrain will be applied to four muscle which are . Tender point of each muscle will be identified then the muscle will be positioned passively in the most relaxed position which will be held for 90 sec. This procedure will repeated 3 times for each muscle
  Other Names: Positional Release
  Arms: Strain-counterstrain Group A
Procedure: Muscle Energy Technique — Muscle energy technique will be applied to four muscles which are quadratus Lumborum, iliacus, piriform and erector spinae. Each muscle will be positioned passively in stretched position the patient asked to push against the therapist isometrically while holding breath for 5-10sec. After exhalation, the muscle will be moved into a new barrier. This procedure will repeated 3 times for each muscle
  Arms: Muscle Energy Technique Group B

SUMMARY:
Examine the effect of strain-counter strain (SCS) versus muscle energy technique (MET) on pain pressure threshold (PPT), functional disability, and the innominate angle tilt with SIJ dysfunction.

DETAILED DESCRIPTION:
Sacroiliac joint dysfunction (SIJD) can be cured with medical and physical therapy interventions. Standard physical therapy techniques include manual joint mobilization, manipulation, bracing, massage, patient education, aerobic training, general exercise, and electrotherapies such as heat, ultrasound, and transcutaneous electric nerve stimulation(TENS). In the physiotherapy context, an effective treatment strategy for unappreciated SIJD is needed. Currently, there are no guidelines or appropriate management plans for this dysfunction, physicians usually refer to it as low back pain alone, and physiotherapists treat the pain as low back pain (LBP). However, appropriate medical intervention or physical therapy may be carried out if the diagnosis is accurate. Furthermore, only a few studies tried to compare the effects of the various treatment approaches.

Strain-counterstain (SCS) consider an excellent choice for building patient thrust as the patient is held passively in a pain-free position. SCS can facilitate treatment for the patient who has experienced pain during a treatment session by using other manual therapy techniques such as manipulation and MET or specific core stability exercises to enhance force closure of SIJ.

SCS allows normalization of the tone of tight muscles involved in SIJ dysfunction which allows a significant improvement in recruitment of weak muscles, especially the gluteal group. SCS has shown its effectiveness in reducing pain or palpation tenderness over different musculoskeletal disorders such as acute/ chronic LBP, mechanical neck pain, and masseter trigger points.

SCS affects local circulations which lead to more nutrient supply, metabolic waste removal, and reverse ischemia that can manifest as painful tender points (TPs) or sustain dysfunction. Current literature lacks consensus on mechanisms, contributing factors, and treatment of SIJ dysfunction.

MET was advocated for the treatment of muscle imbalances in the lumbopelvic region, such as pelvic asymmetry. The theory behind MET assumes that the technique is used to correct asymmetry by targeting hamstring or hip flexor contractions on the painful side of the lower back and move the innominate in the proper direction. It is important to note, however, that evidence indicates that non-symptomatic individuals have also been shown to have pelvic asymmetries.

While manual therapy is a helpful tool for LBP care, few studies have focused on the efficacy of SIJD. There is limited evidence concerning the efficacy of SCS and MET in SIJ dysfunction. According to investigators' knowledge, there is no study to investigate the effectiveness of SCS on SIJ dysfunction patients in comparison to muscle energy technique.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged from 20 years to 60 years.
2. Positive Fortin's sign (pain around PSIS and sacral sulcus).
3. Positive three posterior provocation tests of four including Thigh thrust test, Compression test, Distraction Test, and Patrick test.
4. Pain in lower back below level L5 vertebra and buttocks.
5. Self-reported disability due to SIJ pain on the Oswestry Disability Index (ODI) scores at least 30%.

Exclusion Criteria:

1. Acute injury or fracture of the lower limb and spine.
2. Systemic diseases such as Rheumatoid arthritis (R.A) or ankylosing spondylitis.
3. Previous major lumbar or hip surgery.
4. Pregnancy or delivery for less than 6 months ago.
5. Lumbar stenosis or spondylolisthesis or disc disease.
6. Congenital spinal deformity.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2020-08-08 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Pain Pressure Threshold(PPT) via Digital Pressure Algometer (Wagner Model FDIX) | 10 minutes
  The algometry (Wagner model FDIX) is an analogue mechanical pressure dynamometer with half circular compression rubber tip (1 cm²). The dial ranges from 2.0 to 20.0 kg (kilogram-force). The value of the kilogram-force is equal to a kilogram per square centimeter. PPT will be considered abnormal when it is equal to 3.0 kg or less Two measure points will be marked 2 cm cranially (first point) and 2 cm laterally (second point) from reference point located 1 cm medially and caudally from the posterior superior iliac spine (PSIS) which shows the most painful points in SIJ patients. Anatomically, the first point is related to the attachment of gluteus maximus to the iliac crest while the second point is related to the erector spinae muscle and posterior sacroiliac ligament.
Pelvic tilting via Palpation Meter (PALM) | 15 minutes
  Palpation Meter (PALM) was developed to measure pelvic torsion, pelvic tilting and leg length discrepancy (LLD). The body of the PALM contains a bubble level in a semi-circular arc with one-degree gradations that range from zero degree to thirty degrees on either side of the midline. The caliper arms are placed in bony landmarks and the degree of deviation from horizontal is read from the inclinometer

SECONDARY OUTCOMES:
Functional disability via the Oswestry Disability Index ( ODI): | 15 minutes
  Oswestry Disability Index (ODI) ODI is a validated and well-accepted measure of disability due to lower back pain without distinguishing between different causes of back pain. ODI focused on details of LBP concerning standing, walking, sitting, lifting, daily activity and socially. It is consists of ten questions, each question has a score between 0 and 5.
  The scoring is calculated by dividing total score by the maximum score and multiplied by 100 to give a percentage which indicates the level of disability related to spinal disorder ( 0-20% minimal, 20%-40% moderate, 40%-60% severe, 60%-80% crippled and 80%-100% patient are confined to bed)

CONTACTS AND LOCATIONS:
Overall Officials: Bassem G El- Nahaas, Professor, Study Director
Locations (1):
- Warraq Central hospital, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No